CLINICAL TRIAL: NCT02737202
Title: Safety and Efficacy of Saracatinib In Subjects With Lymphangioleiomyomatosis
Acronym: SLAM-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Cincinnati (Other); Brigham and Women's Hospital (Other); Stanford University (Other); Loyola University (Other); University of South Florida (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nicola Hanania, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLAM 7602; 4UH3TR000961-02 (NIH)
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Lymphangioleiomyomatosis
Keywords: LAM
MeSH Terms: interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Saracatinib (Experimental): Saracatinib will be given orally at a dose of 125 milligrams once daily for 9 months. Saracatinib is provided as a pink tablet.
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib — Subjects will receive enough tablets for 90 days +/- 14 days at each visit. Subject will have visits every 90 days for drug accountability as well as safety and efficacy testing to include pulmonary function testing, laboratory testing to include liver and kidney profile, urine pregnancy testing at each visit, vital signs, physical examination - any medically significant changes from baseline visit will be recorded, all adverse events will be monitored until resolution.
  Other Names: AZD0530

SUMMARY:
This study is being done to determine if there is a potential benefit of saracatinib in LAM subjects. Based on the information of this trial, additional clinical development trials will be needed. The study will also test the tolerability of 125 mg of saracatinib given once daily over a 9 month period.

DETAILED DESCRIPTION:
Tuberous sclerosis complex (TSC) is an autosomal dominant disorder caused by mutations in tuberous sclerosis complex 1 (TSC1) or TSC2 tumor suppressor genes. TSC is characterized by tumors in a wide range of tissues, seizures, mental retardation, autism, and organ failure. Lymphangioleiomyomatosis (LAM), the major pulmonary manifestation in women with TSC, is a progressive lung disease characterized by infiltration of atypical smooth muscle like cells (TSC-/- LAM cells) and formation of parenchymal cysts. Sporadic LAM can develop in women who do not meet the criteria for the diagnosis of TSC, owing to somatic mutations in the TSC2 gene.

The long term goal of this research is to devise novel therapeutic strategies for patients with LAM. The observed behavior of LAM cells with respect to their infiltrative growth pattern, metastatic potential, and altered cell differentiation is reminiscent of cells undergoing epithelial-mesenchymal transition (EMT). Src kinases are key regulators of cellular proliferation, motility, invasiveness and EMT. Recent results have shown that autophagy promotes degradation of active Src. Thereby, decreased autophagy due to mTOR activation known to occur in LAM cells, may play a significant role in accumulation of active Src in these cells. Src suppresses transcription of E-cadherin by upregulating its transcriptional repressors. The preliminary data reveal an increase in active Src in lung tissues of patients with LAM as well as in cultured TSC2-/- cells. Further, in TSC2-/- cells, E-cadherin is considerably reduced and does not localize to the plasma membrane, as it does in wild-type cells.

The focus of this study is to examine if Src inhibition represents a potential therapeutic strategy in LAM. It is proposed that Src activation in TSC2-/- cells results in the reduction of E-cadherin, loss of cell-cell adhesion and elevation of oncogenic and metastatic potential of these cells. The increased Src activity in TSC2-/- cells is likely caused by inhibition of autophagy associated with hyper-activation of mTOR. Therefore, the use of Src inhibitors may lead to a reduction in tumor growth and prevent dissemination of TSC2-/- cells. In this study, the investigators will evaluate the safety and efficacy of Src inhibition in subjects with LAM.

A number of inhibitors of Src are now in clinical trials in patients with a range of different tumors. Dasatinib, an oral adenosine triphosphate (ATP)-competitive Src inhibitor, is now approved for clinical use in patients with chronic myeloid leukemia or acute lymphoblastic leukemia. However, dasatinib has wider 'off target' inhibitory activity than saracatinib including potent activity against Abl, ephrin receptor kinases, platelet-derived growth factor receptor and c-KIT (type of receptor tyrosine kinase and a type of tumor marker. Also called CD117 and stem cell factor receptor.) In contrast, saracatinib has a >10-fold preference for Src over Abl kinases and has very little activity against other tyrosine and serine/threonine kinases. Saracatinib has been already characterized in multiple clinical trials in terms of safety and pharmacokinetics.

The investigators have conducted a Phase1b study to test the safety of various doses of Saracatinib in LAM subjects. The purpose of the Phase1b trial was to determine the optimal dose in terms of safety and tolerability in LAM population. Three escalating doses of saracatinib; 50, 125 and 175 mg were studied. Saracatinib was given orally once a day. Overall, subjects tolerated Saracatinib well. The investigators chose the dose of 125 mg to conduct further testing of both safety and efficacy in this Phase 2a trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients. It should be noted that LAM occurs almost exclusively in women.
* 18 to 65 years of age.
* All patients must have a diagnosis of LAM as defined by compatible cystic changes on chest computed tomography (CT) and one of the following:
* Open lung, transbronchial or thoracic needle biopsy consistent with LAM
* Open or needle abdominal biopsy findings consistent with LAM
* Clinical findings of tuberous scleroma complex (TSC), renal angiomyolipoma, cystic abdominal lymphangiomas, or history of chylous effusion in the chest or abdomen
* Serum vascular endothelial growth factor D (VEGF-D) > 800 pg/ml
* Subjects must have had a recent reduction in forced expiratory volume at 1-second (FEV1) of > 50ml/year, as shown by at least two pulmonary function testing (PFT) measured at least 6 months apart in the last 24 months prior to enrolling study.

Exclusion Criteria:

* Current infection.
* Major surgery within the past 2 months
* Advanced hematologic, renal, hepatic, non-LAM lung disease or metabolic diseases; or BMI of >35
* The use of another investigational drug within 30 days
* The use of mTOR (mammalian target of rapamycin) inhibitors within 30 days
* Previous lung transplantation.
* Inability to attend scheduled clinic visits
* Inability to give informed consent
* Inability to perform pulmonary function testing
* History of malignancy in the past two years, other than squamous or basal cell skin cancer or status post successful excision or treatment.
* Nursing mothers
* Current or planned pregnancy.
* Not using adequate contraception (in woman of childbearing potential).
* Significant clinical change in health in the past 30 days

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
FEV1 | 9 months

SECONDARY OUTCOMES:
Angiomyolipoma measured volumetrically on MRI | 12 months
Lung Cyst size measured on chest CT | 9 months
VEGF-D serum levels | 12 months

OTHER OUTCOMES:
Pulmonary Function Testing | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tony Eissa, MD, Study Chair — Baylor College of Medicine; Nicola A Hanania, MD, Principal Investigator — Ben Taub Hospital; Francis X McCormack, MD, Principal Investigator — University of Cincinnati; Daniel Dilling, MD, Principal Investigator — Loyola University; Stephen Ruoss, MD, Principal Investigator — Stanford University; Joel Moss, MD, Principal Investigator — Laboratory of Translational Research - NHLBI
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Loyola Medical Center, Chicago, Illinois
  - Laboratory of Translational Research NHLBI, Bethesda, Maryland
  - University of Cincinnati, Cincinnati, Ohio
  - Baylor College of Medicine - Ben Taub General Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young J, Povey S. The genetic basis of tuberous sclerosis. Mol Med Today. 1998 Jul;4(7):313-9. doi: 10.1016/s1357-4310(98)01245-3. PMID 9743993
- [Background] Kobayashi T, Minowa O, Sugitani Y, Takai S, Mitani H, Kobayashi E, Noda T, Hino O. A germ-line Tsc1 mutation causes tumor development and embryonic lethality that are similar, but not identical to, those caused by Tsc2 mutation in mice. Proc Natl Acad Sci U S A. 2001 Jul 17;98(15):8762-7. doi: 10.1073/pnas.151033798. Epub 2001 Jul 3. PMID 11438694
- [Background] Kwiatkowski DJ. Tuberous sclerosis: from tubers to mTOR. Ann Hum Genet. 2003 Jan;67(Pt 1):87-96. doi: 10.1046/j.1469-1809.2003.00012.x. PMID 12556239
- [Background] European Chromosome 16 Tuberous Sclerosis Consortium. Identification and characterization of the tuberous sclerosis gene on chromosome 16. Cell. 1993 Dec 31;75(7):1305-15. doi: 10.1016/0092-8674(93)90618-z. PMID 8269512
- [Background] van Slegtenhorst M, de Hoogt R, Hermans C, Nellist M, Janssen B, Verhoef S, Lindhout D, van den Ouweland A, Halley D, Young J, Burley M, Jeremiah S, Woodward K, Nahmias J, Fox M, Ekong R, Osborne J, Wolfe J, Povey S, Snell RG, Cheadle JP, Jones AC, Tachataki M, Ravine D, Sampson JR, Reeve MP, Richardson P, Wilmer F, Munro C, Hawkins TL, Sepp T, Ali JB, Ward S, Green AJ, Yates JR, Kwiatkowska J, Henske EP, Short MP, Haines JH, Jozwiak S, Kwiatkowski DJ. Identification of the tuberous sclerosis gene TSC1 on chromosome 9q34. Science. 1997 Aug 8;277(5327):805-8. doi: 10.1126/science.277.5327.805. PMID 9242607
- [Background] Costello LC, Hartman TE, Ryu JH. High frequency of pulmonary lymphangioleiomyomatosis in women with tuberous sclerosis complex. Mayo Clin Proc. 2000 Jun;75(6):591-4. doi: 10.4065/75.6.591. PMID 10852420
- [Background] Franz DN, Brody A, Meyer C, Leonard J, Chuck G, Dabora S, Sethuraman G, Colby TV, Kwiatkowski DJ, McCormack FX. Mutational and radiographic analysis of pulmonary disease consistent with lymphangioleiomyomatosis and micronodular pneumocyte hyperplasia in women with tuberous sclerosis. Am J Respir Crit Care Med. 2001 Aug 15;164(4):661-8. doi: 10.1164/ajrccm.164.4.2011025. PMID 11520734
- [Background] Astrinidis A, Khare L, Carsillo T, Smolarek T, Au KS, Northrup H, Henske EP. Mutational analysis of the tuberous sclerosis gene TSC2 in patients with pulmonary lymphangioleiomyomatosis. J Med Genet. 2000 Jan;37(1):55-7. doi: 10.1136/jmg.37.1.55. PMID 10633137
- [Background] Illouz F, Braun D, Briet C, Schweizer U, Rodien P. Endocrine side-effects of anti-cancer drugs: thyroid effects of tyrosine kinase inhibitors. Eur J Endocrinol. 2014 Sep;171(3):R91-9. doi: 10.1530/EJE-14-0198. Epub 2014 May 15. PMID 24833135
- [Background] Neelakantan P, Rezvani K, May P, Gerrard G, Marco B, Paliompeis C, Reid A, Goldman J, Marin D, Milojkovic D. Excellent outcome after repeated changes of tyrosine kinase inhibitor therapy for chronic myeloid leukaemia in complete cytogenetic response due to minor side effects. Br J Haematol. 2014 Feb;164(4):608-10. doi: 10.1111/bjh.12648. Epub 2013 Nov 13. No abstract available. PMID 24219400
- [Background] Tyryshkin A, Bhattacharya A, Eissa NT. SRC kinase is a novel therapeutic target in lymphangioleiomyomatosis. Cancer Res. 2014 Apr 1;74(7):1996-2005. doi: 10.1158/0008-5472.CAN-13-1256. PMID 24691995
- [Background] Goncharova EA, Goncharov DA, Damera G, Tliba O, Amrani Y, Panettieri RA Jr, Krymskaya VP. Signal transducer and activator of transcription 3 is required for abnormal proliferation and survival of TSC2-deficient cells: relevance to pulmonary lymphangioleiomyomatosis. Mol Pharmacol. 2009 Oct;76(4):766-77. doi: 10.1124/mol.109.057042. Epub 2009 Jul 13. PMID 19596836
- [Background] Siemann DW, Dong M, Pampo C, Shi W. Src-signaling interference impairs the dissemination of blood-borne tumor cells. Cell Tissue Res. 2012 Aug;349(2):541-50. doi: 10.1007/s00441-012-1415-7. Epub 2012 Apr 18. PMID 22526632
- [Background] Dong M, Rice L, Lepler S, Pampo C, Siemann DW. Impact of the Src inhibitor saracatinib on the metastatic phenotype of a fibrosarcoma (KHT) tumor model. Anticancer Res. 2010 Nov;30(11):4405-13. PMID 21115886
- [Background] Green TP, Fennell M, Whittaker R, Curwen J, Jacobs V, Allen J, Logie A, Hargreaves J, Hickinson DM, Wilkinson RW, Elvin P, Boyer B, Carragher N, Ple PA, Bermingham A, Holdgate GA, Ward WH, Hennequin LF, Davies BR, Costello GF. Preclinical anticancer activity of the potent, oral Src inhibitor AZD0530. Mol Oncol. 2009 Jun;3(3):248-61. doi: 10.1016/j.molonc.2009.01.002. Epub 2009 Feb 7. PMID 19393585
- [Background] Jones RJ, Young O, Renshaw L, Jacobs V, Fennell M, Marshall A, Green TP, Elvin P, Womack C, Clack G, Dixon JM. Src inhibitors in early breast cancer: a methodology, feasibility and variability study. Breast Cancer Res Treat. 2009 Mar;114(2):211-21. doi: 10.1007/s10549-008-9997-1. Epub 2008 Apr 14. PMID 18409068
- [Background] Carsillo T, Astrinidis A, Henske EP. Mutations in the tuberous sclerosis complex gene TSC2 are a cause of sporadic pulmonary lymphangioleiomyomatosis. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6085-90. doi: 10.1073/pnas.97.11.6085. PMID 10823953
- [Background] Dalton RN, Chetty R, Stuart M, Iacona RB, Swaisland A. Effects of the Src inhibitor saracatinib (AZD0530) on renal function in healthy subjects. Anticancer Res. 2010 Jul;30(7):2935-42. PMID 20683035
- [Background] Leeming DJ, Sand JM, Nielsen MJ, Genovese F, Martinez FJ, Hogaboam CM, Han MK, Klickstein LB, Karsdal MA. Serological investigation of the collagen degradation profile of patients with chronic obstructive pulmonary disease or idiopathic pulmonary fibrosis. Biomark Insights. 2012;7:119-26. doi: 10.4137/BMI.S9415. Epub 2012 Sep 13. PMID 23012495
- [Background] Taveira-Dasilva AM, Stylianou MP, Hedin CJ, Hathaway O, Moss J. Bone mineral density in lymphangioleiomyomatosis. Am J Respir Crit Care Med. 2005 Jan 1;171(1):61-7. doi: 10.1164/rccm.200406-701OC. Epub 2004 Oct 1. PMID 15466255
- [Background] Brooks D, Solway S, Gibbons WJ. ATS statement on six-minute walk test. Am J Respir Crit Care Med. 2003 May 1;167(9):1287. doi: 10.1164/ajrccm.167.9.950. No abstract available. PMID 12714344
- [Background] Chapman AB, Guay-Woodford LM, Grantham JJ, Torres VE, Bae KT, Baumgarten DA, Kenney PJ, King BF Jr, Glockner JF, Wetzel LH, Brummer ME, O'Neill WC, Robbin ML, Bennett WM, Klahr S, Hirschman GH, Kimmel PL, Thompson PA, Miller JP; Consortium for Radiologic Imaging Studies of Polycystic Kidney Disease cohort. Renal structure in early autosomal-dominant polycystic kidney disease (ADPKD): The Consortium for Radiologic Imaging Studies of Polycystic Kidney Disease (CRISP) cohort. Kidney Int. 2003 Sep;64(3):1035-45. doi: 10.1046/j.1523-1755.2003.00185.x. PMID 12911554
- [Background] Young LR, Inoue Y, McCormack FX. Diagnostic potential of serum VEGF-D for lymphangioleiomyomatosis. N Engl J Med. 2008 Jan 10;358(2):199-200. doi: 10.1056/NEJMc0707517. No abstract available. PMID 18184970
- [Background] Seyama K, Kumasaka T, Souma S, Sato T, Kurihara M, Mitani K, Tominaga S, Fukuchi Y. Vascular endothelial growth factor-D is increased in serum of patients with lymphangioleiomyomatosis. Lymphat Res Biol. 2006;4(3):143-52. doi: 10.1089/lrb.2006.4.143. PMID 17034294
- [Background] Stacker SA, Caesar C, Baldwin ME, Thornton GE, Williams RA, Prevo R, Jackson DG, Nishikawa S, Kubo H, Achen MG. VEGF-D promotes the metastatic spread of tumor cells via the lymphatics. Nat Med. 2001 Feb;7(2):186-91. doi: 10.1038/84635. PMID 11175849
- [Background] Achen MG, Jeltsch M, Kukk E, Makinen T, Vitali A, Wilks AF, Alitalo K, Stacker SA. Vascular endothelial growth factor D (VEGF-D) is a ligand for the tyrosine kinases VEGF receptor 2 (Flk1) and VEGF receptor 3 (Flt4). Proc Natl Acad Sci U S A. 1998 Jan 20;95(2):548-53. doi: 10.1073/pnas.95.2.548. PMID 9435229
- [Background] Hennequin LF, Allen J, Breed J, Curwen J, Fennell M, Green TP, Lambert-van der Brempt C, Morgentin R, Norman RA, Olivier A, Otterbein L, Ple PA, Warin N, Costello G. N-(5-chloro-1,3-benzodioxol-4-yl)-7-[2-(4-methylpiperazin-1-yl)ethoxy]-5- (tetrahydro-2H-pyran-4-yloxy)quinazolin-4-amine, a novel, highly selective, orally available, dual-specific c-Src/Abl kinase inhibitor. J Med Chem. 2006 Nov 2;49(22):6465-88. doi: 10.1021/jm060434q. PMID 17064066
- [Background] Recchia I, Rucci N, Funari A, Migliaccio S, Taranta A, Longo M, Kneissel M, Susa M, Fabbro D, Teti A. Reduction of c-Src activity by substituted 5,7-diphenyl-pyrrolo[2,3-d]-pyrimidines induces osteoclast apoptosis in vivo and in vitro. Involvement of ERK1/2 pathway. Bone. 2004 Jan;34(1):65-79. doi: 10.1016/j.bone.2003.06.004. PMID 14751564
- [Background] Hannon RA, Clack G, Rimmer M, Swaisland A, Lockton JA, Finkelman RD, Eastell R. Effects of the Src kinase inhibitor saracatinib (AZD0530) on bone turnover in healthy men: a randomized, double-blind, placebo-controlled, multiple-ascending-dose phase I trial. J Bone Miner Res. 2010 Mar;25(3):463-71. doi: 10.1359/jbmr.090830. PMID 19775203
- [Background] de Vries TJ, Mullender MG, van Duin MA, Semeins CM, James N, Green TP, Everts V, Klein-Nulend J. The Src inhibitor AZD0530 reversibly inhibits the formation and activity of human osteoclasts. Mol Cancer Res. 2009 Apr;7(4):476-88. doi: 10.1158/1541-7786.MCR-08-0219. PMID 19372577
- [Background] Baselga J, Cervantes A, Martinelli E, Chirivella I, Hoekman K, Hurwitz HI, Jodrell DI, Hamberg P, Casado E, Elvin P, Swaisland A, Iacona R, Tabernero J. Phase I safety, pharmacokinetics, and inhibition of SRC activity study of saracatinib in patients with solid tumors. Clin Cancer Res. 2010 Oct 1;16(19):4876-83. doi: 10.1158/1078-0432.CCR-10-0748. Epub 2010 Aug 30. PMID 20805299
- [Background] Yu JJ, Robb VA, Morrison TA, Ariazi EA, Karbowniczek M, Astrinidis A, Wang C, Hernandez-Cuebas L, Seeholzer LF, Nicolas E, Hensley H, Jordan VC, Walker CL, Henske EP. Estrogen promotes the survival and pulmonary metastasis of tuberin-null cells. Proc Natl Acad Sci U S A. 2009 Feb 24;106(8):2635-40. doi: 10.1073/pnas.0810790106. Epub 2009 Feb 6. PMID 19202070
- [Background] Goncharova EA, Goncharov DA, Fehrenbach M, Khavin I, Ducka B, Hino O, Colby TV, Merrilees MJ, Haczku A, Albelda SM, Krymskaya VP. Prevention of alveolar destruction and airspace enlargement in a mouse model of pulmonary lymphangioleiomyomatosis (LAM). Sci Transl Med. 2012 Oct 3;4(154):154ra134. doi: 10.1126/scitranslmed.3003840. PMID 23035046
- [Background] Taveira-DaSilva AM, Steagall WK, Moss J. Lymphangioleiomyomatosis. Cancer Control. 2006 Oct;13(4):276-85. doi: 10.1177/107327480601300405. PMID 17075565
- [Background] Puls LN, Eadens M, Messersmith W. Current status of SRC inhibitors in solid tumor malignancies. Oncologist. 2011;16(5):566-78. doi: 10.1634/theoncologist.2010-0408. Epub 2011 Apr 26. PMID 21521831
- [Background] McCormack FX, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Young LR, Kinder BW, Downey GP, Sullivan EJ, Colby TV, McKay RT, Cohen MM, Korbee L, Taveira-DaSilva AM, Lee HS, Krischer JP, Trapnell BC; National Institutes of Health Rare Lung Diseases Consortium; MILES Trial Group. Efficacy and safety of sirolimus in lymphangioleiomyomatosis. N Engl J Med. 2011 Apr 28;364(17):1595-606. doi: 10.1056/NEJMoa1100391. Epub 2011 Mar 16. PMID 21410393
- [Background] Parkhitko A, Myachina F, Morrison TA, Hindi KM, Auricchio N, Karbowniczek M, Wu JJ, Finkel T, Kwiatkowski DJ, Yu JJ, Henske EP. Tumorigenesis in tuberous sclerosis complex is autophagy and p62/sequestosome 1 (SQSTM1)-dependent. Proc Natl Acad Sci U S A. 2011 Jul 26;108(30):12455-60. doi: 10.1073/pnas.1104361108. Epub 2011 Jul 11. PMID 21746920
- [Background] Tyryshkin A, Gorgun FM, Abdel Fattah E, Mazumdar T, Pandit L, Zeng S, Eissa NT. Src kinase-mediated phosphorylation stabilizes inducible nitric-oxide synthase in normal cells and cancer cells. J Biol Chem. 2010 Jan 1;285(1):784-92. doi: 10.1074/jbc.M109.055038. Epub 2009 Oct 29. PMID 19875457
- [Background] Marin TM, Clemente CF, Santos AM, Picardi PK, Pascoal VD, Lopes-Cendes I, Saad MJ, Franchini KG. Shp2 negatively regulates growth in cardiomyocytes by controlling focal adhesion kinase/Src and mTOR pathways. Circ Res. 2008 Oct 10;103(8):813-24. doi: 10.1161/CIRCRESAHA.108.179754. Epub 2008 Aug 28. PMID 18757826